CLINICAL TRIAL: NCT07391605
Title: A RANDOMIZED DOUBLE-BLIND PLACEBO-CONTROLLED STUDY TO EVALUATE EFFICACY, SAFETY, AND TOLERABILITY OF DESCARTES-08 IN PATIENTS WITH DERMATOMYOSITIS AND ANTISYNTHETASE SYNDROME
Brief Title: Descartes-08 in Autoantibody Myositis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cartesian Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RNAC-TRITON-08
Record Dates: First submitted 2026-01-29; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Antisynthetase Syndrome
Keywords: MYOSITIS; DESCARTES-08; MRNA CAR-T; TOTAL IMPROVEMENT SCORES; CDASI
MeSH Terms: conditions — Antisynthetase syndrome; Myositis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Decartes-08 (Experimental)
  Interventions: Drug: Descartes-08
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Descartes-08 — Autologous T-cells expressing a chimeric antigen receptor (CAR) directed to B-Cell maturation antigen (BCMA)
  Arms: Decartes-08
Other: Placebo — Plasma-Lyte
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase 2 study to evaluate the efficacy, safety and tolerability of an autologous T-cells expressing a chimeric antigen receptor (CAR) directed to B-Cell maturation antigen (BCMA) in patients with autoantibody-mediated myositis, including antisynthetase syndrome (ASyS) and dermatomyositis (DM).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of one of the following:

Dermatomyositis (DM): Probability score ≥55% on the 2017 EULAR/ACR (European Alliance of Associations of Rheumatology/ American College of Rheumatology) criteria for classification of dermatomyositis (corresponding to diagnosis of 'probable or definite' DM). OR Antisynthetase Syndrome (ASyS): Diagnosis based on ACR/EULAR Classification Criteria (1)."

* Participants must have dermatomyositis or antisynthetase syndrome with muscle and/or skin involvement.
* Refractory or intolerance to standard therapy.
* Stable background immunosuppressive therapy for ≥8 weeks.
* Adequate hematologic, renal, hepatic, and pulmonary function (SpO₂ ≥92% on room air).
* Informed consent, compliance with visits, contraception, and vaccinations required.

Exclusion Criteria:

* Isolated interstitial lung disease (ILD) without muscle or skin involvement

  * Severe irreversible muscle damage or advanced weakness (e.g., wheelchair-bound).
  * Interstitial lung disease (ILD) requiring oxygen, severe pulmonary impairment (FVC ≤45%, DLCO ≤40%), or pulmonary hypertension.
  * Other inflammatory myopathies (PM, IMNM, IBM, cancer- or drug-induced myositis, overlap myositis except Sjögren's).
  * Other severe neuromuscular, cardiac, pulmonary, or systemic autoimmune diseases requiring immunosuppression.
  * Significant uncontrolled chronic illnesses or psychiatric conditions interfering with participation.
  * Pregnancy or lactation.
  * Recent use of prohibited immunosuppressants/biologics or investigational agents (per washout periods).
  * Live vaccination within 4 weeks.
  * History of primary immunodeficiency, organ or bone marrow transplant.
  * Active or uncontrolled infections: HBV, HCV, HIV, tuberculosis, or recurrent/severe infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Major improvement of 2016 ACR/EULAR Total Improvement score | 24 weeks
  Proportion of participants in the Descartes-08 group compared with placebo who achieve major improvement marked by ≥60 point improvement on the 2016 ACR/EULAR Total Improvement Score (TIS)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fedak, R.R., Ruggerie, R.N., Shan, Y. et al. BCMA-directed mRNA CAR-T cell therapy for myasthenia gravis: exploratory biomarker analysis of a placebo-controlled phase 2b trial. Nat Med (2026). https://doi.org/10.1038/s41591-025-04170-z
- See also: Related Info — https://rdcu.be/e1nFI